CLINICAL TRIAL: NCT00608829
Title: Evaluation of the GORE TAG® Thoracic Endoprosthesis - 45 mm for the Primary Treatment of Aneurysms of the Descending Thoracic Aorta
Brief Title: GORE TAG® Thoracic Endoprosthesis - 45 mm for the Treatment of Aneurysms of the Descending Thoracic Aorta
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: W.L.Gore & Associates (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAG 06-02
Record Dates: First submitted 2007-12-20; First posted 2008-02-06 (Estimated); Results first posted 2010-09-15 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2015-03

CONDITIONS: Aortic Aneurysm, Thoracic
MeSH Terms: conditions — Aortic Aneurysm, Thoracic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GORE TAG® Thoracic Endoprosthesis (Experimental): Gore 45mm TAG Thoracic Endograft Implantation
  Interventions: Device: GORE TAG® Thoracic Endoprosthesis

INTERVENTIONS:
Device: GORE TAG® Thoracic Endoprosthesis — Implant
  Other Names: GORE TAG® Thoracic Endoprosthesis - 45 mm

SUMMARY:
The objective of this study is to assess the safety and efficacy of the 45 mm TAG device in subjects with aneurysms of the descending thoracic aorta.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of Descending thoracic aortic aneurysm deemed to warrant surgical repair

   * Fusiform (≥50 mm), or
   * Saccular (no diameter criteria)
2. All proximal and/or all distal landing zone inner diameters between 37-42 mm

   * Diameter taper between proximal and distal landing zones and the ability to use devices of different diameters to compensate for the taper must be within device sizing guide specifications
3. Proximal and distal landing zone length greater than 2.0 cm

   * Landing zone must not be aneurysmal, dissected, heavily calcified, or heavily thrombosed
4. Life expectancy > 2 years
5. Subject is open surgical candidate defined as:

   * Able to tolerate thoracotomy
   * American Society of Anesthesiologists class I-IV (class V excluded)
   * New York Heart Association class I-III or not applicable (class IV excluded)
6. Male or infertile female
7. Age greater than 21 years
8. Able to comply with study protocol requirements, including follow-up

Exclusion Criteria:

1. Mycotic aneurysm
2. Hemodynamically unstable aneurysm rupture
3. Aortic dissection
4. Planned occlusion of left carotid or celiac arteries
5. Planned concomitant surgical procedure (other than left subclavian transposition), or major surgery within 30 days of treatment date
6. Myocardial infarction or stroke within 6 weeks of treatment
7. Pre-treatment creatinine > 2.0 mg/dL
8. Degenerative connective tissue disease, e.g. Marfan's or Ehler-Danlos Syndrome
9. Participation in another drug or device study within 1 year of treatment
10. History of drug abuse within 6 months of treatment

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2007-02; Primary Completion 2009-08 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michel Makaroun, MD, Principal Investigator — University of Pittsburgh Medical Center
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- 45mm TAG Device Subjects: The TAG device is a flexible, self-expanding stent graft used for endovascular repair of the Descending Thoracic Aorta. The 45 mm TAG device is a true "line extension", as it is identical to the approved 26-40 mm GORE TAG Thoracic Endoprosthesis, with the exception of the diameter.
Period: Overall Study
Arm/Group | 45mm TAG Device Subjects
Started | 23
Completed | 8
Not Completed | 15
Not completed — Death | 6
Not completed — Withdrawal by Subject | 4
Not completed — Subject refuses to follow up or return. | 5

BASELINE CHARACTERISTICS:
Arm/Group | 45mm TAG Device Subjects
Number analyzed (Participants) | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 77.6 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 19
Region of Enrollment [Number; unit: participants]
  United States | 23

OUTCOME MEASURES:

1. Primary Outcome: Freedom From Major Adverse Events and Major Device Events Through 1 Year Post-treatment
Description: Major Adverse Event: a) requires therapy and short hospitalization (24 - 48 hours), b) requires major therapy, unplanned increase in level of care, prolonged hospitalization (>48 hours), c) permanent adverse sequelae, or d) death. (Sacks et. al.; JVIR, 1997; 8:137-149).
Time Frame: one year
Measure: Number; unit: Participants
Arm/Group | 45mm TAG Device Subjects
Number analyzed (Participants) | 23
Participants | 11

ADVERSE EVENTS:
Time Frame: Up to 5 years of follow-up
Description: Note: Major/Minor classification was collected. All events classified as 'Major' are in 'Serious adverse events', 'Minor' events are in 'Other adverse events'. Major adverse events were those resulting in: a)therapy and short hospitalization b)major therapy/increase in level of care/prolonged hospitalization c)permanent adverse sequelae or d)death.
Arm/Group | 45mm TAG Device Subjects
Serious Adverse Events (participants affected / at risk) | 17/23
Other Adverse Events (participants affected / at risk) | 19/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 45mm TAG Device Subjects (N=23)
Bleeding Complication (Blood and lymphatic system disorders) | 5
Cardiac Complication (Cardiac disorders) | 6
Bowel Complication (Gastrointestinal disorders) | 2
Sepsis (Infections and infestations) | 2
Endoleak (Injury, poisoning and procedural complications) | 3
Wound Complication (Injury, poisoning and procedural complications) | 2
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neurologic Complication (Nervous system disorders) | 4
Genitourinary (Renal and urinary disorders) | 2
Renal Function Complication (Renal and urinary disorders) | 3
Pulmonary Complication (Respiratory, thoracic and mediastinal disorders) | 5
Other Complication (Social circumstances) | 8
Vascular Complication (Vascular disorders) | 5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 45mm TAG Device Subjects (N=23)
Bleeding Complication (Blood and lymphatic system disorders) | 5
Cardiac Complication (Cardiac disorders) | 8
Bowel Complication (Gastrointestinal disorders) | 3
Endoleak (Injury, poisoning and procedural complications) | 10
Wound Complication (Injury, poisoning and procedural complications) | 2
Neurologic Complication (Nervous system disorders) | 5
Genitourinary (Renal and urinary disorders) | 3
Renal Function Complication (Renal and urinary disorders) | 4
Pulmonary Complication (Respiratory, thoracic and mediastinal disorders) | 9
Other Complication (Social circumstances) | 12
Vascular Complication (Vascular disorders) | 2

LIMITATIONS AND CAVEATS:
Enrollment into this trial was completed prematurely with 23 enrolled subjects. The 45mm TAG Device was approved based on the data collected and a descriptive statistical analysis. Follow up of enrolled subjects continued for 5 years.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Gore has the right to review disclosures, requesting a delay of more than 60 days but less than or equal to 180 days. Each investigator will postpone single center publications until after disclosure of multi-center data, less than 12 months from study completion/termination at all participating sites.